CLINICAL TRIAL: NCT02796040
Title: Exploration of Mesocorticolimbic Pathway in Impulse Control Disorders in Parkinson's Disease: Study Using Tensor Diffusion Imaging and Tractography.
Acronym: TCI-IRMdiff
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0266
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Parkinson's Disease; Impulse Control Disorders
Keywords: Parkinson's disease; Impulse control disorders; Diffusion tensor imaging; MRI; Mesocorticolimbic pathway
MeSH Terms: conditions — Parkinson Disease; Disruptive, Impulse Control, and Conduct Disorders

ARMS (2):
- patients with ICD (impulse control disorder) (Experimental): More precisely, the main purpose is to demonstrate that fractional anisotropy (FA) (data obtained with DTI) in the ventral tegmental area (VTA) is different between patients with ICD and patients without ICD
  Interventions: Device: MRI
- patients without ICD (impulse control disorder) (Other): More precisely, the main purpose is to demonstrate that fractional anisotropy (FA) (data obtained with DTI) in the ventral tegmental area (VTA) is different between patients with ICD and patients without ICD
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI

SUMMARY:
Impulse control disorders (ICD) are frequent in Parkinson's Disease. Neurobiological substrates of these symptoms are largely unknown.

The investigators aim to explore mesocorticolimbic pathway in Parkinson's disease patients with impulse control disorders (ICD) using an MRI technique called tensor diffusion imaging (DTI).

More precisely, the main purpose is to demonstrate that fractional anisotropy (FA) (data obtained with DTI) in the ventral tegmental area (VTA) is different between patients with ICD and patients without ICD. Secondary objectives are to demonstrate a difference in volume of VTA, in FA in others structures included in reward system (prefrontal cortex, nucleus accumbens, amygdala), and in number of fibers between VTA and the other structures of reward system between this two groups. Other objective is to measure and compare these same variables between Parkinson's patients and healthy controls.

We hypothesized that a denervation of mesocorticolimbic pathway predisposes Parkinson's patients to ICD.

DETAILED DESCRIPTION:
Type of study: Prospective, case control study.

Number of centers: 1 (Clermont-Ferrand)

Patients :

Inclusion of 25 patients with Parkinson's disease and impulse control disorders (inclusion's criteria detailed later), 25 matched Parkinson's disease patients without impulse control disorders and 25 healthy volunteers.

Study Performance :

J0 (inclusion; 3 hours) :

Each subject will perform a clinical and neurological examination (UPDRS) and a neuropsychological evaluation for diagnostic and quantification of impulse control disorders and to ensure of the absence of exclusion criteria.

J0+1week (MRI; 1hour) Each subject will then have an MRI acquisition including anatomical sequences (T1 and T2 weighted sequences) and a diffusion tensor imaging sequence (60 directions).

Analysis Analysis (Pre-processing and processing) will be realized with the Oxford Centre for Functional MRI of the Brain (FMRIB) Software (FSL).

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease (UK Parkinson's Disease Society Brain Bank Criteria)
* from 18 to 85 years old
* Impulse control disorder (one item ICD ≥2 at the scale ECMP : Evaluation Comportementale de la maladie de Parkinson)

Exclusion Criteria:

* Dementia (Mini Mental State < 26 or MATTIS < 130)
* Apathy (LARS (Lille Apathy Rating Scale) > 7)
* Depression (MADRS (Montgomery and Alsberg Depression Scale) ≥16
* Contra indication to MRI (claustrophobia, deep brain stimulation, pace maker…)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Fractional anisotropy (data of diffusion tensor imaging, a technique of MRI) | 1 day

SECONDARY OUTCOMES:
Fractional anisotropy in préfrontal cortex | 1 day
Volume of ventral tegmental area | 1 day
Number of fibers between ventral tegmental area and other structures of the reward system | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Franck DURIF, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France